CLINICAL TRIAL: NCT02908542
Title: Search for New Genetic Causes of Hypercalcemia by Massively Parallel Sequencing of a Genes Panel
Acronym: HyCaGene
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-048
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2016-09

CONDITIONS: Hypercalcemia
MeSH Terms: conditions — Hypercalcemia | interventions — Genetic Testing; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood or DNA samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: genetic analysis with massively parallel sequencing

SUMMARY:
Hypercalcemia, whether chronic or acute, exposes the patient to potentially serious complications (arrhythmias, nephrolithiasis, nephrocalcinosis, ...). Prevention relies primarily on effective etiological necessary for taking matched load. Under the French reference center for rare disorders of calcium and phosphorus, the investigators looked for mutations in the coding sequence of the CYP24A1 gene (encoding the enzyme responsible for the breakdown of vitamin D), among patients with hypercalcemia without hyperparathyroidism with hypersensitivity to vitamin D. However, only 25% of these patients have a genetic anomaly suggesting the involvement of other genes (Molin et al. 2015). Recently our team, combined with Kaufmann et al. (2014 JCEM) validated the interest of the determination of metabolites of vitamin D by liquid chromatography-tandem mass spectrometry (LC-MS / MS), as biological pre-screening stage for patients with hypercalcemia.

The objective of this project is to complement the molecular and biochemical studies of patients without mutation of the coding sequence of CYP24A1, in a gene candidate approach using massively parallel sequencing (MPS) which allows to study a panel of gene potentially involved in disorder of metabolism of calcium and phosphorus. Highlighted variations will be tested in silico, and if possible in vitro. The investigators will also use LC-MS / MS to evaluate in vivo the effects of these variations on the metabolism of vitamin D, to develop a genotype / phenotype correlation.

The work carried out within the Genetics Department Caen University Hospital in collaboration with physicians of the rare disease reference center of the metabolism of calcium and phosphorus should identify new genetic mechanisms underlying hypercalcemia. At the time of development of personalized medicine, it will adapt the therapy in patients at risk for metabolic complications and / or kidney following administration of vitamin D and finally to offer genetic counseling.

ELIGIBILITY:
Inclusion criteria

* Chronic hypercalcemia or at least one episode of acute hypercalcemia not linked to hyperparathyroidism
* Consent to the realization of a genetic analysis for medical purposes Non-inclusion criteria
* Another genetic disorder identified with hypercalcemia (eg Williams-Beuren syndrome)
* Primary hyperparathyroidism (high PTH)
* neoplasia
* granulomatosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with medical history of hypercalcemia without hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-12; Primary Completion 2017-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
number of identified genetic variations presumed pathogenic | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Caen Hospital University, Caen, France

IPD SHARING:
Plan to Share IPD: Yes
The data will be communicated to the referent physician of the patient.